CLINICAL TRIAL: NCT00069056
Title: A Pilot Study of Laser Photocoagulation for Diabetic Macular Edema
Brief Title: Pilot Study of Laser Photocoagulation Therapy for Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030291; 03-EI-0291
Record Dates: First submitted 2003-09-13; First posted 2003-09-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Diabetic Retinopathy
Keywords: Grid Laser; Focal Laser; Glycemic Control; Diabetes; Diabetic Macular Edema; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Macular Edema | interventions — Laser Therapy

INTERVENTIONS:
Procedure: Laser Treatment

SUMMARY:
This study will compare the side effects of two laser treatments for diabetic macular edema, a common condition in patients with diabetes. In macular edema, blood vessels in the retina, a thin layer of tissue that lines the back of the eye, become leaky and the retina swells. The macula, the center part of the retina that is responsible for fine vision, may also swell and cause vision loss. Traditional laser treatment (argon blue or green, or yellow) for macular swelling, or edema, causes scarring that can expand and possibly lead to more loss of vision. A different laser technique, the mild macular grid, uses lighter laser burns through the macula and may be less damaging to the eye, but this is not known. This study will compare the two techniques and the information on side effects will be used to design a larger study of whether one laser is more effective than the other.

Patients 18 years of age and older with type 1 or type 2 diabetes and macular edema may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history and physical examination.
* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils will be dilated with drops for this examination.
* Blood tests to measure cholesterol levels, hemoglobin A1C (a measure of diabetes control), and creatinine (measure of kidney function).
* Eye photography to help evaluate the status of the retina and changes that may occur in the future. Special photographs of the inside of the eye are taken using a camera that flashes a bright light into the eye.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Optical coherence tomography to examine retinal thickness. The eye is examined with a machine that produces cross-sectional pictures of the retina. These measurements will be repeated during the study to determine whether retinal thickening is getting better, worse, or staying the same.

Participants will be randomly assigned to one of the two laser therapies in the eye with macula edema. (Patients with macular edema in both eyes will receive both treatments-one in each eye.) For these procedures, eye drops are put in the eye to numb the surface, and a contact lens is placed on the eye during the laser beam application. Several visits may be required for additional laser treatments. The number of treatments depends on how well they are working. Patients will return for follow-up visits 4, 8, and 12 months after the first treatment, and then every year until year 3. During the follow-up visits, the response to treatment will be evaluated with repeat tests of several of the screening exams.

DETAILED DESCRIPTION:
The Diabetic Retinopathy Clinical Research Network (DRCRnet) was formed to conduct clinical trials and epidemiological studies for diabetic retinopathy.

As part of the establishment of the network, it is necessary to standardize data collection methods, testing procedures, and treatment techniques for use in the anticipated multiple protocols to be conducted by the network. One of the treatment techniques requiring standardization is laser photocoagulation treatment of diabetic macular edema. To accomplish this goal, a protocol has been developed to enroll patients with diabetic macular edema who require laser treatment. Procedures to be conducted by standardized protocols include refraction, visual acuity testing, fundus photography, fluorescein angiography, optical coherence tomography (OCT) and laser photocoagulation. One of the benefits from having a structured protocol will be that the outcome data using the standardized techniques can be used for sample size estimations in future protocols. This is particularly true for OCT for which we need to develop standard methods to assess changes in groups of patients and for which there are limited longitudinal data, especially in groups of patients.

The conduct of this study provides the opportunity not only to collect data on a standardized laser protocol commonly used in current clinical practice but also to collect pilot data evaluating a new laser technique. The 'current practice' laser protocol, modified from the ETDRS treatment protocol, involves focal/grid photocoagulation to areas of macular thickening with leaking MA, diffuse leakage or nonperfusion (modified-ETDRS technique). There is extensive evidence supporting the efficacy of ETDRS laser photocoagulation technique for the treatment of macular edema. The alternative technique, called mild macular grid (MMG) photocoagulation, provides mild grid treatment using small, widely separated burns to the retina from 500 to 3000 microns (3500 microns temporally) from the macular center. This technique may potentially have fewer side effects, different edema resolution rate or prevention of future development of macular edema as discussed below. The study will use randomization to assign each patient to receive one of the two treatment methods.

For this protocol, participation will be open to all clinical sites that have the requisite equipment needed for the study and to all ophthalmologists who meet criteria to be a DRCR.net investigator. The sample size for the study will be dictated by the number of participating sites, with each site limited to the enrollment of a maximum of four patients or one patient per certified investigator, whichever is greater.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA - SUBJECT-LEVEL:

  1. Age greater than or equal to 18 years.
  2. Diagnosis of diabetes mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

     1. Current regular use of insulin for the treatment of diabetes.
     2. Current regular use of oral antihyperglycemia agents for the treatment of diabetes.
     3. Documented diabetes by ADA guidelines.
  3. No history of renal failure requiring dialysis or renal transplant.
  4. No condition that in the opinion of the investigator would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control). Patients in poor glycemic control who recently initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 3 months should not be enrolled.
  5. Ability and willingness to provide informed consent.
  6. No expectation that subject will be moving out of the area of the clinical center to an area not covered by another clinical center during the next 12 months.

INCLUSION AND EXCLUSION CRITERIA - STUDY EYE:

At least one eye must meet all of the following criteria:

1. Best corrected ETDRS visual acuity score greater than or equal to 19 letters (approximately 20/400 or better).
2. Definite retinal thickening due to diabetic macular edema based on clinical exam at or within 500 microns of the macular center for which the investigator believes laser photocoagulation is indicated.
3. A thickness of 250 microns or more in the central subfield OR a thickness of 300 microns or more in any one of the four subfields directly adjacent to the central subfield on OCT.
4. No prior focal/grid laser photocoagulation in the macula.
5. No prior medical treatment for DME (e.g., intravitreal/peribulbar steroids).
6. No panretinal scatter photocoagulation (PRP) within prior 4 months.
7. No anticipated need for PRP within next 4 months.
8. No major ocular surgery (including cataract extraction, any other intraocular surgery, scleral buckle, glaucoma filter, cornea transplant, etc.) within prior 6 months.
9. No Nd:YAG laser capsulotomy within prior 2 months.
10. Macular edema is not considered to be due to a cause other than diabetic macular edema. An eye should not be considered eligible (1) if the macular edema is considered to be related to cataract extraction or (2) clinical exam and/or OCT suggests that vitreoretinal interface disease (eg. vitreo-retinal traction or epriretinal membrane) is the primary cause of the macular edema.
11. Media clarity, papillary dilation, and patient cooperation sufficient for adequate fundus photos.
12. No ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the first 12 months of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome). Glaucoma per se is not an exclusion.

A patient may have two "study eyes" only if both are eligible at the time of randomization. An eye that becomes eligible after randomization will not be considered a study eye for purposes of data analyses or treatment decisions although information is being gathered on all eyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4
Dates: Start 2003-09-10; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Diabetic Retinopathy Clinical Research Network, Bethesda, Maryland

REFERENCES:
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759